CLINICAL TRIAL: NCT05708937
Title: Assistant Proffessor Ph.D.
Brief Title: THE EFFECT OF COGNITIVE AWARENESS SUPPORT ON THE PSYCHOSOCIAL STATUS OF WOMEN TREATED FOR INFERTILITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Özen İnam, Lecturer, Maltepe University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-74555795-050.01.04-52289
Record Dates: First submitted 2022-12-19; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Infertility; Infertility, Female
Keywords: Infertility; Female Infertility; Mindfulness
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group participants used the mindfulness mobile application. Then, the psychosocial status of the participants was measured with scales.
  Interventions: Behavioral: Mindfulness based phone app
- Control group (No Intervention): The control group participants did not receive any intervention. Classical care was applied. Then, the psychosocial status of the participants was measured with scales.

INTERVENTIONS:
Behavioral: Mindfulness based phone app — Creating mindfulness-based suggestions for infertile women:
  Mindfulness-based content was created by taking the opinions of experts in the fields of women's health nursing, psychology and linguistics. It consists of 6 different parts. The content of meditation that the patient will apply according to the treatment stage is different. Infertility mindfulness departments; "Breath Awareness, Body & Uterus Awareness, Needle Therapy and Ovarian Awareness, Pre-Egg Collection (OPU) Diaphragm Breathing, Pre-embryo Transfer Uterine Awareness, Embryo and Uterine Awareness (Post transfer)".
  Audio recordings of mindfulness-themed meditation content:
  After the meditation contents are planned; the sound recording was taken with a professional recorder (Sony ICD-PX470). The audio recordings taken were professionally edited by the expert. Mp3 recordings were created by adding background music to sound recordings in computer environment. Audio recordings of mindfulness-themed meditation content
  Arms: Experimental group

SUMMARY:
Aim: With the project, mobile application supported cognitive awareness applications in women receiving infertility treatment; The aim of this study was to measure the effect of infertile women on their psychosocial status.

Method: It was planned as a randomized controlled study. It was aimed to reduce stress and increase awareness by applying mindfulness/cognitive awareness to women undergoing infertility treatment. For this reason, special mindfulness suggestions were created for infertile women by taking the opinion of an expert in the field. Mindfulness suggestions created specifically for women with infertility were recorded. The recordings were varied according to the treatment stages, with an average duration of 40 minutes. These audio recordings were presented with a mobile application developed for infertile women. The mobile application called IVFMind was designed for infertile women. The application consists of mindfulness audio recordings and reading sections. The experimental group (n:17) installed this application on their phones and listened to the audio recordings regularly. Cognitive awareness (BIFO), depression-anxiety (DASS 21), infertility self-efficacy and fertility adjustment scales were administered to the experimental and control groups (N:34). Scales were done as pre-test and post-test. The mobile application evaluation form was filled in the experimental group.

DETAILED DESCRIPTION:
Infertility is a process with social, cultural and psychological interaction as well as physical condition. Infertility is a perceived loss for women, men and families. It requires adapting to a childless lifestyle and developing a coping mechanism with the difficulties encountered (Lee, Choi, Chan , Chan , & Ernest, 2009). Infertility treatments are stressful, physically painful and financially demanding life crises for most couples (Boivin, Griffiths, & Venetis, 2011). It is not enough that the nursing care that women who experience such a complex psychosocial process will receive during the same complex treatment process is only physical care. For this reason, individuals in the diagnosis and treatment process of infertility, especially women, need social support (Blevins, 2011).

Providing psychosocial support to infertile patients is one of the important tasks of nursing care.

There are studies in the literature showing that mindfulness-based care is an effective method for improving psychological health (such as quality of life, stress, marital adjustment) in women in infertility clinics (Fard, Kalantarkousheh, & Faramarzi, 2018) (Lunn & Sherratt, 2013) (Shargh, et al. , 2016) (Hosseini, et al., 2020). A study of the mindfulness-based care intervention found increases in awareness levels, self-compassion, and coping strategies in infertile women during their first IVF treatment. Thus, it was found to improve fertility-related quality of life and pregnancy rates (Li, Long, Liu, He, & Li, 2016).

With this project, a mobile application was developed to provide mindfulness-based psychosocial support to infertile women. The mobile application contains mindfulness-based audio recordings developed specifically for infertility. Participants listened regularly (twice a day) to meditation appropriate to the treatment phase.

Psychosocial assessments (pretest and posttest) were applied to measure the benefit of this practice on participants.

The psychosocial status of women receiving infertility treatment was measured through the scales used, and the effect of mobile application and mindfulness nursing support on the participants was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having completed the Informed consent form and volunteering to participate in the study
* Not having a psychiatric diagnosis (schizophrenia, bipolar disorder, major depression, anxiety disorders, etc.)
* Beginning or soon to start IVF treatment (starting ovarian stimulation)
* Having a maximum of three previous IVF attempts
* Using a smartphone
* Speaks and understands Turkish
* Being over 18 years old

Exclusion Criteria:

* Termination of treatment at any stage
* Failure to transfer embryos
* Leaving work voluntarily

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 6 weeks
  This form, prepared by the researcher, consists of 21 items. It questions socio-demographic information such as age, educational status, occupation, duration of marriage, and infertility history, obstetric history and chronic disease status.
Cognitive Awareness Scale | 1 year
  Developed by Brown and Ryan in 2003, the scale aims to measure awareness and attention to momentary experiences in daily life. It gives the total score with its single factor structure, as the score increases, the level of conscious awareness increases. Factor loads range from 27 to 78. It is answered on a 15-item 6-point Likert-type scale (from "almost always" to "almost never"). It aims to determine how often they experience their experiences automatically, without paying attention to the present moment. As the scores obtained from the scale increase; It is understood that cognitive awareness is high. The internal consistency coefficient of the scale is 82
Infertility Self-Efficacy Scale | 1 year
  The original titled Infertility Self-Efficacy Scale was found in 2006 by Cousineau et al. It was developed to evaluate the self-efficacy perceptions of individuals related to infertility about their emotional, cognitive and behavioral skills.
  The nine-point Likert-type scale (1- not at all important and 9- very important) consists of a total of 16 items. In 2006, a 10-item short form was created. All statements in the scale are positive. Scores ranging from 10 to 90 are taken from the short form of the scale. The higher the score, the higher the perception of self-efficacy. In the original of the scale, the reliability coefficient was determined as α:94. The scale is unidimensional and scores are between 8 and 32. The higher the score, the higher the perception of self-efficacy.
Depression Anxiety Stress Short Scale (DASS 21) | 1 year
  Depression anxiety stress short scale (DASS 21) consists of 21 items aiming to measure the level of "depression, anxiety and stress" under three headings. In the normal sample, the test-retest correlation coefficients were found to be r=0.68 for the depression subscale, r=0.66 for the anxiety subscale, and r=0.61 for the stress subscale. This scale is a 4-point Likert-type scale and measures "depression, stress and anxiety dimensions". If the individual scores 5 points or more from the depression sub-dimension, 4 points or more from anxiety, and 8 points or more from stress, it indicates that he or she has a related problem.
Mobile Application Evaluation Results | 1 year
  It was prepared by the researcher and aims to evaluate users' satisfaction with the mobile application. The usability of the mobile application is aimed at getting the opinions of the patients about the topics to be suggested for the mobile application. The first 4 items of the 6-item form have a 3-point Likert feature (1-yes, 2-no, 3-I'm not sure), while the other 2 items ask open-ended questions about the topics that users want to suggest.
Fertility Adjustment Scale | 1 year
  The scale, originally named Fertility Adjustment, was developed by Glover et al in 1999 to standardize the measurement of psychological adjustment in infertility. Infertility compliance; It is considered as a concept that includes behavioral, cognitive and emotional aspects. The infertility adjustment scale can be used as a useful tool to evaluate the effect of the treatment process on the psychosocial adjustment of individuals and their psychological needs. The scale is a six-point Likert-type, 12-item scale. The minimum scale score is 12 and the maximum score is 72. The items were balanced in order not to affect the answers in terms of positive and negative statements. Positive items are reverse scored. A high infertility compliance scale score indicates inadequate compliance. In the original of the scale, the reliability coefficient was determined as α.85.

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe Üniversitesi, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Inam O, Satilmis IG. The effect of mindfulness-based nursing support on the psychosocial status of women receiving infertility treatment: a randomized controlled trial. BMC Womens Health. 2025 Mar 20;25(1):127. doi: 10.1186/s12905-025-03659-6. PMID 40114156